CLINICAL TRIAL: NCT06993181
Title: An Open-label, Randomized, Fasting, Single-dose, 2-sequence, 2-period, Crossover Phase 1 Study to Compare and Evaluate the Pharmacokinetic Characteristics and the Safety After Single-administration of DA-5222 and Co-administration of DA-5222-R1, DA-5222-R2 and DA-5222-R3 in Healthy Adult Subjects
Brief Title: Clinical Trial of Comparing DA-5222 Single-administration and Co-administration of DA-5222-R1, DA-5222-R2 and DA-5222-R3 in Healthy Adult Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA5222_BE_I
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: DA-5222, DA-5222-R1, DA-5222-R2, DA-5222-R3
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: DA-5222; Drug: DA-5222-R1; Drug: DA-5222-R2; Drug: DA-5222-R3
- Sequence B (Experimental)
  Interventions: Drug: DA-5222; Drug: DA-5222-R1; Drug: DA-5222-R2; Drug: DA-5222-R3

INTERVENTIONS:
Drug: DA-5222 — single dose administration (DA-5222 one tablet once a day)
Drug: DA-5222-R1 — single dose administration (DA-5222-R1 one tablet once a day)
Drug: DA-5222-R2 — single dose administration (DA-5222-R2 one tablet once a day)
Drug: DA-5222-R3 — single dose administration (DA-5222-R3 one tablet once a day)

SUMMARY:
This study is to compare pharmacokinetics and safety profiles of DA-5222 single-administration and co-administration of DA-5222-R1, DA-5222-R2 and DA-5222-R3 in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI between 18 and 30 kg/m2
* Body weight: Male≥50kg, Female≥45kg
* Subjects who have signed an informed consent themselves after receiving detailed explanation about clinical study

Exclusion Criteria:

* Subjects with clinically significant medical history
* Subjects with history of drug abuse or addicted
* Subjects with allergy or drug hypersensitivity

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
AUCt | pre-dose~72 hours post-dose
  area under the curve
Cmax | pre-dose~72 hours post-dose
  maximum plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Bumin Hospital, Seoul, South Korea, South Korea